CLINICAL TRIAL: NCT02466139
Title: Early Clinical, Laboratory and Microbiological Predictors of Treatment Outcomes Among Infective Endocaridtis Patients in a Tertiary-care Centre in Kerala
Brief Title: Early Clinical, Laboratory and Microbiological Predictors of Treatment Outcomes in Infective Endocaridtis
Acronym: CRP-IE
Status: Completed | Type: Observational
Sponsor: Government Medical College, Kozhikode (Other)
Responsible Party: Principal Investigator, Sandeep Mohanan, Senior Resident (DM) Cardiology, Government Medical College, Kozhikode
Other Study IDs: IEregister2012-2015
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Infective Endocarditis
Keywords: microbiology; c reactive protein; urgent cardiac surgery
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators conduct a prospective observational study on consecutive patients being admitted to a tertiary care-centre with infective endocarditis. The investigators' primary aim is to identify baseline clincal, laboratory and microbiological predictors of in-hospital events, mortality and 6-month mortality.

DETAILED DESCRIPTION:
Mortality and major complications among infective endocarditis remain high. In addition developing nations are crippled with a high incidence of culture-negative endocarditis and lack of wide availability of transesophageal echocardiography. We intended to identify predictors among admission clinical features, laboratory paramters and culture reports that can help risk stratify patients early in the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of modified Duke criteria

Exclusion Criteria:

* No consent
* inadequate baseline data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with infective endocarditis treated in a tertiary care centre
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days
Major complications | 30 days

SECONDARY OUTCOMES:
Number of patients who had embolic events | 30 days
Number of patients who needed urgent cardiac surgery | 30 days
Short term Mortality | 6 months